CLINICAL TRIAL: NCT00579644
Title: Treatment of Early Rheumatoid Arthritis: Minocycline in Combination With Methotrexate Versus Methotrexate Alone
Brief Title: Treatment of Early RA: Minocycline in Combination With Methotrexate vs Methotrexate Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0519-00 FB
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 Methotrexate* & minocycline (Active Comparator): Methotrexate Dosing:
  1)initial dose of methotrexate for all patients will be 10 mg/week. 2)2 month: dose of MTX will remain at 10 mg/week if full remission criteria are met; otherwise, increased to 15 mg/week.
  3)4 month: dose of MTX will remain at its current level if full remission criteria are met; otherwise, be increased to 20 mg/week.
  4)6, 8 and 10 month: If the patient has fallen below full remission criteria and is not already receiving the maximum dose of 20 mg/week,dose will be increased to 20 mg/week. If the patient meets ACR 50 criteria prednisone will be tapered by 1mg/month 5)12 month evaluation: End of the blinded portion of the study. minocycline dosage 200 mg
  Interventions: Drug: Combination of Minocycline and MTX or MTX alone
- 2 Methotrexate (Active Comparator): Methotrexate Dosing:
  1. Initial evaluation: The dose of methotrexate for all patients will be 10 mg/week.
  2. 2 month evaluation: The dose of MTX will remain at 10 mg/week if full remission criteria are met; otherwise, it will be increased to 15 mg/week.
  3. 4 month evaluation: The dose of MTX will remain at its current level if full remission criteria are met; otherwise, it will be increased to 20 mg/week.
  4. 6, 8 and 10 month evaluations:
     * If the patient has fallen below full remission criteria and is not already receiving the maximum dose of 20 mg/week, the dose will be increased to 20 mg/week.
     * If the patient meets ACR 50 criteria prednisone will be tapered by 1mg/month
  5. 12 month evaluation: End of the blinded portion of the study.
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: Combination of Minocycline and MTX or MTX alone — Methotrexate Dosing:
  1)initial dose of methotrexate for all patients will be 10 mg/week. 2)2 month: dose of MTX will remain at 10 mg/week if full remission criteria are met; otherwise, increased to 15 mg/week.
  3)4 month: dose of MTX will remain at its current level if full remission criteria are met; otherwise, be increased to 20 mg/week.
  4)6, 8 and 10 month: If the patient has fallen below full remission criteria and is not already receiving the maximum dose of 20 mg/week,dose will be increased to 20 mg/week. If the patient meets ACR 50 criteria prednisone will be tapered by 1mg/month 5)12 month evaluation: End of the blinded portion of the study. minocycline dosage 200 mg
  Other Names: Rheumatrex®; Trexall®; Dynacin®; Minocin®; Myrac®
  Arms: 1 Methotrexate* & minocycline
Drug: methotrexate — Initial evaluation: The dose of methotrexate for all patients will be 10 mg/week.
  2 month evaluation: The dose of MTX will remain at 10 mg/week if full remission criteria are met; otherwise, it will be increased to 15 mg/week.
  4 month evaluation: The dose of MTX will remain at its current level if full remission criteria are met; otherwise, it will be increased to 20 mg/week.
  6, 8 and 10 month evaluations:
  If the patient has fallen below full remission criteria and is not already receiving the maximum dose of 20 mg/week, the dose will be increased to 20 mg/week.
  If the patient meets ACR 50 criteria prednisone will be tapered by 1mg/month 12 month evaluation: End of the blinded portion of the study.
  Other Names: Rheumatrex®; Trexall®
  Arms: 2 Methotrexate

SUMMARY:
The purpose of this study is to determine if a combination of methotrexate and minocycline works better than methotrexate alone in early Rheumatoid Arthritis

DETAILED DESCRIPTION:
The purpose of this study is to determine if a combination of methotrexate and minocycline works better than methotrexate alone in early Rheumatoid Arthritis (RA). Specific aims of this study are:

A. To demonstrate that the combination of minocycline and methotrexate is well tolerated when used in the first year of RA.

B. To compare the efficacy of the combination of minocycline and methotrexate with methotrexate and placebo therapy in early sero-positive RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over or equal to 19 years old and less than or equal to 75 years old
* Diagnosis of RA as determined by fulfilling 4 of 7 ACR criteria
* Positive rheumatoid factor
* Duration of disease: greater than six weeks and less than one year

Exclusion Criteria:

* Allergy to tetracycline or methotrexate
* Previous DMARD treatment
* Doses of oral steroids greater than 7.5 mg/day
* Intra-articular injections within the last four weeks
* Significant liver or renal disease or active peptic ulcer disease
* Patients who are not willing to abstain from alcohol consumption
* Women of childbearing potential who are not practicing a successful method of contraception

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2001-03-28 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2006-05-31 (Actual)

PRIMARY OUTCOMES:
Remission evaluated by American College of Rheumatology (ACR) outcome variables | 48 weeks
  Patients will be evaluated and then at 2-month intervals to 12 months using the ACR core set of outcome variables (50) for remission. Additionally hand x-rays will be done.

SECONDARY OUTCOMES:
Comparison of combination therapy versus methotrexate alone, Composite Index | 48 weeks
  Clinically relevant comparison of the effectiveness of combination therapy versus methotrexate alone will be improvement by 20% and/or 70% by the American College of Rheumatology composite index.

CONTACTS AND LOCATIONS:
Overall Officials: James R O'Dell, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States